CLINICAL TRIAL: NCT06235736
Title: Do Patients With Anterior Cruciate Ligament (ACL) Tears Demonstrate Weakness of the Soleus Muscle?
Brief Title: Do Patients With ACL Tears Demonstrate Weakness of the Soleus Muscle?
Acronym: ACL
Status: Recruiting | Type: Observational
Sponsor: University of Liverpool (Other)
Responsible Party: Sponsor
Other Study IDs: UoL001827
Record Dates: First submitted 2024-01-23; First posted 2024-02-01 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: ACL Tear; ACL-injury; ACL - Anterior Cruciate Ligament Rupture
Keywords: Acute cruciate ligament; ACL; soleus muscle; physiotherapy; orthopaedics; trauma; rehabilitation
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Wounds and Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MRI-confirmed ACL tear group: This group will have had a complete ACL tear confirmed by MRI scan
- Normative group: This group will provide normative data for the study. They will have no previous history of significant knee injury and no current symptomatic lower limb injuries.

SUMMARY:
The goal of this prospective, cross-sectional study is to test the strength of the soleus muscle in participants who have a ACL tear confirmed by MRI. Previous studies have shown that the soleus muscle, which one of the muscles situated in the calf, decreases mechanical loading on the ACL. Therefore, we aim to test soleus muscle strength using a seated plantar flexor test.

The main questions we aim to answer are:

* Do patients with ACL tears demonstrate inter-limb soleus strength asymmetry (>10%)
* Do patients with ACL tears have soleus muscle weakness compared with uninjured (normative) participants?
* Do changes in soleus strength values correlate with patient reported outcomes and stability, as measured by the IKDC questionnaire?

To achieve this the VALD force frame will be used as the testing device for plantar flexor strength testing. This device records the force generated by the movement. This will be repeated three times on each leg as part of the testing procedure. Furthermore, as part of the testing procedure participants will be required to fill out an IKDC form to assess their knee stability. Interrater reliability of the force frame will be investigated.

Further data from participants without ACL tears will be used to compare results. Thus allowing us to see if people with ACL tears have a weakness in the soleus muscle.

DETAILED DESCRIPTION:
To address the research question, we will collect and analyse measures of lower limb muscle strength, which together will inform on the strength/ weakness of the Soleus muscle in patients undergoing physiotherapy rehabilitation following MRI-confirmed ACL injury.

Patients identified as eligible according to the protocol inclusion and exclusion criteria will be invited to participate in the study through informed written consent so that their clinical measurements can be used as research data. Healthy volunteers will be identified by direct email invitation or word of mouth. Healthy volunteers will be members of staff at Aintree Hospital, LUHFT.

Patients will undergo the clinically established treatment pathway for rehabilitation with lower limb muscle strength and performance measurements taken from isometric seated calf raise using the Vald Forceframe and single leg jump using Vald Forcedecks. Measurements will be performed with maximal ankle dorsiflexion and the knee flexion angle greater than 90 degrees. Three submaximal warmups will be performed followed by three maximum efforts, taking the maximum reading for analysis.

Normative values from healthy participants will be collected using the same clinical protocol.

Patients and healthy participants will be asked to complete the international knee documentation committee (IKDC) questionnaire at the start and end of rehabilitation, to determine subjective complaints of instability.

ELIGIBILITY:
Inclusion Criteria:

ACL tear participants:

* MRI-confirmed ACL tear.
* Participant is willing and able to give informed consent in writing for participation in the study.
* Male or Female, aged 18 years to 55 years of age.
* No contraindications to strength testing (see exclusion criteria).

Normative values from healthy individuals:

* No current or previous history of significant lower limb injury, or a history of previous minor injury that is symptomatic at the time of recruitment.
* No previous lower limb surgery.
* No course of medication, whether prescribed or over the counter, other than vitamins and mineral supplements or, for females, oral contraceptives.

Exclusion Criteria:

* History of chronic musculoskeletal disease or disorder in either leg that may put the participants at risk because of participation in the study including non-united fractures, epilepsy, cardiac insufficiency, severe peripheral vascular disease, aneurysms, anticoagulant therapy, recent (<3 months) radiotherapy or chemotherapy, long term steroid use (>3 months), pregnancy, neurological disorders (e.g., Parkinson's disease), skin conditions at point of force testing, severe osteoporosis, malignancy, rheumatoid arthritis.

  * Conditions or symptoms that may influence the result of the study, or the participant's ability to participate in the study including pain, limited range of motion, knee effusion, or anaemia.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A convenience sample of MRI-confirmed ACL injured patients, who are undergoing non-operative rehabilitation, will be recruited from Liverpool University Hospitals NHS Trust.. To account for potential bilateral weakness in muscle strength, normative values from a control group of healthy participants will be included. Healthy volunteers will be recruited from NHS staff at Liverpool University Hospitals NHS Foundation Trust. Volunteers will be approached directly via departmental email and face to face conversation or accepted via word of mouth. The international knee documentation committee (IKDC) questionnaire will be completed by the patient, to determine subjective knee stability.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2024-01-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Force generated | 30 minutes
  The primary outcome will be to measure the force generated by the soleus muscle in both limbs. This data will be normalised to their body weight to compare.

SECONDARY OUTCOMES:
IKDC score | 5 minutes
  Participants will be required or complete an IKDC score to assess their knee stability

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Oldershaw, Principal Investigator — University of Liverpool
Locations (1):
- Aintree Hospital, Liverpool University Hospitals NHS Foundation Trust, Liverpool, United Kingdom